CLINICAL TRIAL: NCT00917631
Title: Co-Bedding as a Comfort Measure for Twins Undergoing Painful Procedures
Acronym: CComforT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Marsha Campbell-Yeo, Neonatal Nurse Practitioner, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #4382
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Neonatal Procedural Pain Response
Keywords: Co-bedding; Procedural pain; Twin; Comfort; RCT
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Co-bedding (Experimental): Twin infants will be placed together in a Incubator or crib lying side-by-side. Twins will be diaper clad and nested together in boundaries consistent with neonatal care practices. All infants will have cardio-respiratory monitoring while co-bedding.
  Infants in the co-bedding group be co-bedded for no less than 24 hours prior to heelstick to allow for stabilization following transfer. The heelstick being studied will occur no greater than 10 days following initiation of co-bedding. Duration of co-bedding will be recorded and controlled for in the analysis if necessary.
  Monitoring and video-tape recording will take approximately 20-30 minutes per participant - a baseline period (5-10 minutes prior to heel stick), warming (3 minutes), heel stick (2-5 minutes), and recovery phase (approximately 10 minutes).
  Interventions: Procedure: Co-bedding (caring for twins in the same incubator)
- Standard care (No Intervention): For infants who are randomized to receive standard care, the twin pair will remain in separate incubators as per current NICU policy. The infant will be nested in boundaries consistent with neonatal care practices. The heelstick may occur at any time following randomization (within 10 days) to maintain consistency between groups.

INTERVENTIONS:
Procedure: Co-bedding (caring for twins in the same incubator) — Twin infants will be placed together in a Incubator or crib lying side-by-side. Twins will be diaper clad and nested together in boundaries consistent with neonatal care practices. All infants will have cardio-respiratory monitoring while co-bedding.
  Infants in the co-bedding group be co-bedded for no less than 24 hours prior to heelstick to allow for stabilization following transfer. The heelstick being studied will occur no greater than 10 days following initiation of co-bedding. Duration of co-bedding will be recorded and controlled for in the analysis if necessary.
  Monitoring and video-tape recording will take approximately 20-30 minutes per participant - a baseline period (5-10 minutes prior to heel stick), warming (3 minutes), heel stick (2-5 minutes), and recovery phase (approximately 10 minutes).
  Arms: Co-bedding

SUMMARY:
A rising number of preterm twins, at high risk of undergoing repeated medical procedures often without adequate pain relief, are being admitted to Neonatal Intensive Care Units. Skin-to-skin contact between mothers and their infants during painful procedures has been shown to decrease pain and help them stabilize more quickly afterwards. The main question of this study is whether the contact of a twin could provide a similar form of comfort. Sixty-four twin pairs will have an equal chance of undergoing a medically necessary heel stick while being cared for together (co-bedding) or separately. Primary outcome will be physiologic and behavioral pain response. If found to be beneficial, changes to neonatal care practices to include co-bedding may help twins tolerate and recover from painful procedures. Findings will help care providers make recommendations for at risk twins experiencing procedural pain and add to existing theoretical models with respect to the exact mechanism of comfort through touch.

ELIGIBILITY:
Inclusion Criteria:

* All medically stable twin infants admitted to the NICU who are:

  1. Free from infection; and
  2. Breathing room air or receiving oxygen via nasal prongs.
* Twins may be receiving feeds via gavage tubes, IV therapy via peripheral or central line, and may be experiencing periods of apnea.

Exclusion Criteria:

* Weigh less than 1000 grams;
* Receiving ventilator support;
* Have chest tubes or umbilical catheter in situ;
* Have major congenital anomalies or chromosomal aberrations; OR
* If only one of the twins require overhead phototherapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2008-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Pain response(Premature Infant Pain Profile (PIPP) | Baseline until completion of heelstick

SECONDARY OUTCOMES:
Recovery | The length of time for heart rate and oxygen saturation to return to normal (baseline).
Vagal tone | Baseline until completion of heelstick
Hormonal stress response (Cortisol) | Baseline and 20 minutes post heelstick
Frequency of 24% sucrose administration | Baseline to completion of the heelstick
The response of the co-twin not receiving the painful procedure | Baseline to completion of the heelstick

CONTACTS AND LOCATIONS:
Overall Officials: Marsha L Campbell-Yeo, MN NNP-BC PhDc, Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Campbell-Yeo ML, Johnston CC, Joseph KS, Feeley N, Chambers CT, Barrington KJ, Walker CD. Co-bedding between preterm twins attenuates stress response after heel lance: results of a randomized trial. Clin J Pain. 2014 Jul;30(7):598-604. doi: 10.1097/AJP.0000000000000015. PMID 24300226
- [Derived] Campbell-Yeo ML, Johnston CC, Joseph KS, Feeley N, Chambers CT, Barrington KJ. Cobedding and recovery time after heel lance in preterm twins: results of a randomized trial. Pediatrics. 2012 Sep;130(3):500-6. doi: 10.1542/peds.2012-0010. Epub 2012 Aug 27. PMID 22926182
- [Derived] Campbell-Yeo ML, Johnston CC, Joseph K, Feeley NL, Chambers CT, Barrington KJ. Co-bedding as a Comfort measure For Twins undergoing painful procedures (CComForT Trial). BMC Pediatr. 2009 Dec 11;9:76. doi: 10.1186/1471-2431-9-76. PMID 20003351